CLINICAL TRIAL: NCT00629369
Title: Duration of Second Stage of Labor Wearing a Dental Occlusion Device: a Randomized Controlled Trial
Brief Title: Duration of Second Stage of Labor Wearing a Dental Occlusion Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Robert O. Atlas, MD, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMC2007-39
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): subjects with Occlusion Support Device with active pushing in the second stage of labor
  Interventions: Device: Extra 3 mouth guard, Shock doctor mouth guard v3.0
- 2 (No Intervention): Subjects without Occlusal Support Device with active pushing in the second stage of labor

INTERVENTIONS:
Device: Extra 3 mouth guard, Shock doctor mouth guard v3.0 — Dental mouthguard, molded for each individual patient when in labor. The device is put in the water then in microwave for one minute to soften the device. The device is then applied to the patient's mouth for over 10 seconds to mold it.
  Other Names: extra 3 mouth guard (www.shieldsports.com); shock doctor mouth guard v3.0 (www.shockdoc.com)
  Arms: A

SUMMARY:
Developing a method to maximize maternal expulsive effort should be of great value in reducing the number of cesarean section or instrumental deliveries. Various investigations have shown that use of an occlusal support device (OSD) increases the isometric strength of different muscle groups. The aim of our study was to investigate the role of an OSD in second stage pushing.

DETAILED DESCRIPTION:
The increased use of epidural anesthesia during labor has lead to an increased incidence of prolonged second stage as an indication for cesarean section or instrumental delivery. The use of oxytocin has proven to be an effective method of augmentation of labor in such prolonged labor cases. However, despite oxytocin augmentation, there has been an increase in the number of cases that require cesarean section or instrumental delivery to effect delivery.

McRobert's maneuver, which is often used in to relieve shoulder dystocia, has recently been shown to increase intrauterine pressure approximately two-fold. However; it is an arduous position for the pregnant woman to maintain over a long period of time. Developing alternative methods to maximize expulsive forces, both uterine contractions and maternal expulsive effort, may be of great value in reducing the number of cesarean sections or instrumental deliveries.

Various researchers have investigated the effect of an occlusal support device (OSD) on the isometric strength of different muscle groups, e.g., neck, back, and extremities. The natural condition of dental occlusion, also known as the index of physical performance, has an affect on both muscle strength and body balance. When occlusal support is given to edentulous individuals they show improved physical exercise ability after the re-establishment of mandibular support. Patients whose dentition is in proper occlusion demonstrate greater endurance of isometric muscle strength than those who are in malocclusion. We hypothesize that optimization of dental occlusion by an OSD may improve muscle strength, leading to increased intrauterine pressure during the second stage in labor.

The aim of our study is to investigate whether the use of the OSD results in a shortened duration of the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Primipara
* Term
* Singleton
* Cephalic presentation
* Reactive fetal heart rate pattern
* Functioning epidural anesthesia

Exclusion Criteria:

* Medical or obstetrical complications including intrauterine growth restriction
* Large for gestational age
* Uterine anomaly
* Uterine myomata
* Pre-eclampsia
* Diabetes mellitus
* Fetal anomaly
* Maternal heart disease

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The duration of the second stage of labor. | The duration of the second stage of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Atlas, MD, Principal Investigator — Mercy Medical Center, Baltimore
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Matsuo K, Mudd JV, Kopelman JN, Atlas RO. Duration of the second stage of labor while wearing a dental support device: a pilot study. J Obstet Gynaecol Res. 2009 Aug;35(4):672-8. doi: 10.1111/j.1447-0756.2008.01010.x. PMID 19751326